CLINICAL TRIAL: NCT00256438
Title: The Treatment of Depression Using Transcranial Direct Current Stimulation (tDCS): a Pilot Study.
Brief Title: Depression and Transcranial Direct Current Stimulation (tDCS)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of New South Wales (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05125
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2006-07-10 (Estimated); Status verified 2006-07

CONDITIONS: Depression
Keywords: Depression; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Depression | interventions — Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation

SUMMARY:
Transcranial direct current stimulation (tDCS)is a non invasive technique which uses a very weak current to change excitability in targeted regions of the brain. Early studies suggest that it has antidepressant properties. This study will test the safety and efficacy of tDCS as a treatment for depression.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) applies a weak direct current across the scalp that can produce sub-threshold changes in the excitability of targeted cortical regions, in a polarity-specific manner. This technique has been used in humans to alter motor and visual cortex excitability, during stimulation, and for a period after the stimulation has ceased. It has therefore been suggested as a possible treatment for depression (Lippold & Redfearn, 1964; Nitsche, 2002). Studies have been launched recently to examine the effect of tDCS in depressed subjects and a sham-controlled pilot study (in USA, in press) has reported promising antidepressant effects with tDCS.

We wish to examine this in an investigation of 20 subjects, and hypothesise that tDCS will have an antidepressant effect and produce no neuropsychological impairment. Subjects will receive anodal DC stimulation or sham stimulation over the left prefrontal cortex in a double-blind, placebo-controlled design over 5 days, and then have daily stimulation up to a maximum of 10 active sessions in total. Outcomes will be formally evaluated by depression rating scales and neuropsychological tests.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Major Depressive Episode of less than or equal to 3 years
* Montgomery-Asberg Depression Rating Scale score of 25 or more
* Aged 18-65
* May or may not be taking antidepressant medication

Exclusion Criteria:

* Not able to give written informed consent
* Failure to respond to ECT in current or past episodes of depression
* On antipsychotic, anticonvulsant or benzodiazepine medication which cannot be withdrawn.
* Significant other Axis I psychiatric disorder e.g schizophrenia, bipolar
* In imminent physical or psychological danger and needs a rapid clinical response due to inanition, psychosis or high suicidality
* Drug or alcohol dependence or abuse currently or in the last 12 months
* History of neurological illness e.g epilepsy; neurosurgical procedure
* Metal in the cranium, pacemaker, cochlear implant, medication or other electronic device in the body
* Woman of child-bearing age in whom pregnancy cannot be ruled out by B HCG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-02

PRIMARY OUTCOMES:
All measures at baseline and after each 5 treatments:
Montgomery& Asberg Depression Rating Scale
Hamilton Psychiatric Rating Scale for Depression
Clinical Global Impression-Severity
Beck Depression Inventory
Patient Global Impression-Severity

SECONDARY OUTCOMES:
Neuropsychological assessment at baseline and after each 5 treatments:
Rey Auditory Verbal Learning Task
Digit span
Trail Making Test
Controlled Oral Word Association

CONTACTS AND LOCATIONS:
Overall Officials: Perminder P Sachdev, FRANZCP PhD, Principal Investigator — University of NSW; Colleen K Loo, FRANZCP, MD, Principal Investigator — University of NSW
Locations (1):
- Black Dog Institute Building, School of Psychiatry, University of NSW, Sydney, New South Wales, Australia